CLINICAL TRIAL: NCT06110871
Title: "The Effect of Inhaler Lavender, Focus and Music on Women's Pain, Anxiety, in Intrauterine Device Application"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate (Other Government)
Responsible Party: Principal Investigator, Mine Gokduman Keles, Midwifery, Turkish Ministry of Health, Kahramanmaras Provincial Health Directorate
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TurkishHKahramanmaras
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Visual Analog Pain Scale
Keywords: Virtual Reality; Inhaler Lavende; Pain; Anxiety; Intrauterine Device Application
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: In our research, there will be 3 interventions (Group 1 is a focus group, Group 2 is the Group where inhaled kavanta is used, Group 3 will be listened to music) and 1 control group (The group where IIA is applied and receives routine care). .
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: PERSON USING IUD. IT WILL ALWAYS BE THE SAME AND THERE WILL BE ONE PERSON WHO HAS NOTHING TO DO WITH THE RESEARCH.
  THE RESEARCHER WILL HAVE NO INTERVENTION DURING IUD APPLICATION.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Working Group 1(inhaled lavender) (Experimental): In study group 1, 3 drops of lavender oil will be dropped on aromastone and participants will be asked to inhale deeply 10 times. Then, participants will be allowed to inhale lavender oil for a total of 30 minutes in the waiting room where aromastone is located and in the ria application room.
  Interventions: Other: inhaled lavender
- Working Group 2: Focusing (Experimental): After the internet connection is established with the smartphone, you can click on www.youtube.com and watch the "Relaxation Project 1" (SBS VR) video for the image and ask to focus.
  Interventions: Other: Working Group 2: Focusing
- Working Group 3 music (Experimental): You will be able to listen to Turkish classical music for a total of 30 minutes in the RIA application waiting room and RIA application room.
  Interventions: Other: Working Group 3 music
- Control Group (No Intervention): The care and practices will be the same as in routine IUD application.

INTERVENTIONS:
Other: inhaled lavender — They will be asked to inhale deeply 10 times. Then, a total of 30 minutes in the waiting room where aromastone is located and in the IA application room.
  Arms: Working Group 1(inhaled lavender)
Other: Working Group 2: Focusing — During IUD application
  Arms: Working Group 2: Focusing
Other: Working Group 3 music — for a total of 30 minutes
  Other Names: music
  Arms: Working Group 3 music

SUMMARY:
Randomized control is an experimental study. The purpose of this research; To examine the effects of inhaler lavender, focus and music on women's pain and anxi.ety in intrauterine device application.

In the randomized controlled experimental study, data would be obtained using the Numerical Anxiety Rating Scale and the Numerical Pain Rating Scale. 240 women who underwent IUD procedure at the Family Planning Consultancy Polyclinic of a secondary level public hospital in a city center between October and December 2023 were randomly assigned to receive 4 sets of 1 set of Inhaled lavender (60), 1 set of Focusing (60), 1 set of Music ( 60). 1 control group (60) will participate in the study.

DETAILED DESCRIPTION:
The rate of women who want to use Family Planning in the world has reached approximately 1.1 billion in the last twenty years and has shown a significant increase ( WHO, 2020) . In addition, WHO reported that almost half of the pregnancies in developing countries between 2015 and 2019 were unwanted pregnancies (WHO, 2020) , and recommended effective FP counseling and the use of more modern contraceptive methods to prevent this (WHO, 2020) . In Turkey, the Ministry of Health provides individuals with free access to modern FP methods. Despite this, according to the 2018 data of the Turkey Demographic and Health Survey ( Akdemir and Karadeniz 2019), it has been reported that 49% of the FP method uses modern methods and the Intrauterine Device (IUD) is among the most effective modern methods with a rate of 14% (Akdemir and Karadeniz 2019 ). Factors affecting IUD use include; Women's perception of pain during application and the fact that it can be applied in certain centers (Dine et al,2018; Hunter et al, 2020; Hamdamian et al., 2018).

It has been reported in the literature that women perceive pain during IUD application (Akdemir and Karadeniz 2019; Dine et al,2018; Hunter et al, 2020; Hamdamian et al., 2018). Again, studies have reported the use of inhaled lavender, focus, and music to relieve pain and anxiety (Hamdamian et al., 2018; Hathcock et al., 2021; Türkmen et al.,2021) . These results emphasize the need for low-cost and applicable nonpharmacological methods for healthcare professionals during IUD insertion.

No study has been found in the literature examining the effects of inhaler lavender, focus and music on women's pain and anxiety during intrauterine device application. However, in line with the results of the study, it is thought that it will have a positive effect on reducing the pain and anxiety perceived by women during the IUD procedure.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45,
* having IUD applied for the first time,
* being literate in Turkish,
* having no history of cervical surgery,
* having no active mental illness,
* having no pain before IUD application.

Exclusion Criteria:

* Having communication problems,
* visual or auditory disabilities,
* use of misoprostol during the procedure,
* use of painkillers before the IUD application procedure,
* use of medication for anxiety before the procedure.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Intrauterine Device Application women
Enrollment: 240 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale Pain | Procedure (Speculum insertion)
  Numerical Pain Assessment Scale Pain (NADÖ): Numerical Pain Assessment Scale (NADÖ) is used to evaluate the severity of pain. On the numerical rating scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
Numerical Pain Rating Scale Pain | up to 10 minutes (During the Pap smear test)
  Numerical Pain Assessment Scale Pain (NADÖ): Numerical Pain Assessment Scale (NADÖ) is used to evaluate the severity of pain. On the numerical rating scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
Numerical Pain Rating Scale Pain | 15 minutes after the Pap smear test.
  Numerical Pain Assessment Scale Pain (NADÖ): Numerical Pain Assessment Scale (NADÖ) is used to evaluate the severity of pain. On the numerical rating scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
The Verbal Category Scale | Procedure (Speculum insertion)
  The Verbal Category Scale is also called the Simple Descriptive Scale, and this scale is based on the patient choosing the most appropriate word that describes the pain condition. Pain intensity ranges from mild to unbearable. In this scale, the words "mild", "disturbing", "severe", "very severe", "unbearable" were used to describe the intensity of pain (
The Verbal Category Scale | up to 10 minutes (During the Pap smear test)
  The Verbal Category Scale is also called the Simple Descriptive Scale, and this scale is based on the patient choosing the most appropriate word that describes the pain condition. Pain intensity ranges from mild to unbearable. In this scale, the words "mild", "disturbing", "severe", "very severe", "unbearable" were used to describe the intensity of pain (
The Verbal Category Scale | 15 minutes after the Pap smear test.
  The Verbal Category Scale is also called the Simple Descriptive Scale, and this scale is based on the patient choosing the most appropriate word that describes the pain condition. Pain intensity ranges from mild to unbearable. In this scale, the words "mild", "disturbing", "severe", "very severe", "unbearable" were used to describe the intensity of pain (
Numerical Rating Scale for Anxiety (VASA). | 5 minutes
  Numerical Rating Scale for Anxiety (VASA). It is expressed as whether the individual feels anxiety (e.g., I have a lot of anxiety = 10) or does not feel anxiety (e.g., I have no anxiety = 0).
Numerical Rating Scale for Anxiety (VASA). | 2 minutes
  Numerical Rating Scale for Anxiety (VASA). It is expressed a Outcome 8s whether the individual feels anxiety (e.g., I have a lot of anxiety = 10) or does not feel anxiety (e.g., I have no anxiety = 0).

CONTACTS AND LOCATIONS:
Locations (1):
- TurkishMoHKahramanmarasPH, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akdemir Y, Karadeniz M. The relationship between pain at IUD insertion and negative perceptions, anxiety and previous mode of delivery. Eur J Contracept Reprod Health Care. 2019 Jun;24(3):240-245. doi: 10.1080/13625187.2019.1610872. Epub 2019 May 16. PMID 31094575
- [Background] Dina B, Peipert LJ, Zhao Q, Peipert JF. Anticipated pain as a predictor of discomfort with intrauterine device placement. Am J Obstet Gynecol. 2018 Feb;218(2):236.e1-236.e9. doi: 10.1016/j.ajog.2017.10.017. Epub 2017 Nov 8. PMID 29079143
- [Background] Hunter TA, Sonalkar S, Schreiber CA, Perriera LK, Sammel MD, Akers AY. Anticipated Pain During Intrauterine Device Insertion. J Pediatr Adolesc Gynecol. 2020 Feb;33(1):27-32. doi: 10.1016/j.jpag.2019.09.007. Epub 2019 Sep 26. PMID 31563628
- [Background] Hamdamian S, Nazarpour S, Simbar M, Hajian S, Mojab F, Talebi A. Effects of aromatherapy with Rosa damascena on nulliparous women's pain and anxiety of labor during first stage of labor. J Integr Med. 2018 Mar;16(2):120-125. doi: 10.1016/j.joim.2018.02.005. Epub 2018 Feb 9. PMID 29526235
- [Background] Wojcik A, Bonk K, Muller WU, Obe G, Streffer C. Do DNA double-strand breaks induced by Alu I lead to development of novel aberrations in the second and third post-treatment mitoses? Radiat Res. 1996 Feb;145(2):119-27. PMID 8606920
- [Background] Turkmen H, Cetinkaya S, Kilic H, Apay E, Karamuftuoglu D, Yoruk S, Ozkirim E. Effect of Focusing on Maryam's Flower During the First Stage of the Labor on the Labor Pain, Labor Duration, and Levels of Comfort and Satisfaction. Clin Nurs Res. 2021 Jul;30(6):780-789. doi: 10.1177/1054773820984911. Epub 2020 Dec 29. PMID 33371726
- [Background] Lee JH. The Effects of Music on Pain: A Meta-Analysis. J Music Ther. 2016 Winter;53(4):430-477. doi: 10.1093/jmt/thw012. Epub 2016 Oct 19. PMID 27760797
- [Background] Toker E, Demirel G, Doganer A, Karakucuk S. Effects of Turkish Classical Music on Postpartum Pain and Anxiety in Cesarean Deliveries: A Randomized Controlled Trial. Altern Ther Health Med. 2021 Jun;27(S1):120-127. PMID 33245708
- See also: Family planning/contraception methods. — https://www.who.int/news-room/fact-sheets/detail/family-planning-contraception
- See also: TNSA. (2018 ). Türkiye Nüfus ve Sağlık Araştırması; 2018 — http://www.sck.gov.tr/wp-content/uploads/2020/08/TNSA2018_ana_Rapor.pdf